CLINICAL TRIAL: NCT04767763
Title: Association of Continuous Veno-venous Hemodiafiltration With Citrate Anticoagulation to Thyroid Function in Critically Ill Patients
Brief Title: Thyroid Function in Critically Ill Patients With Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: 02-0064/07/287
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Secondary Hypothyroidism
Keywords: renal replacement therapy; thyroid hormones; acute kidney injury; intensive care unit
MeSH Terms: conditions — Hypothyroidism; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with Acute Kidney Injury: Patients with acute kidney injury and indications for initiation of continuous renal replacement therapy (CRRT) were included to this study irrespective of their gender, race and age.
  Interventions: Diagnostic Test: Assessment of TSH, fT3, fT4,TRH, TT3, TT4, rT3 in patients with CVVHDF

INTERVENTIONS:
Diagnostic Test: Assessment of TSH, fT3, fT4,TRH, TT3, TT4, rT3 in patients with CVVHDF — blood samples were collected before initiation of CRRT and at 1,2,3,6,9-day following. Last samples were collected 3 days after the end of CRRT.

SUMMARY:
The objective of this study was to assess the changes in thyroid hormones and its activity during CRRT in patients with Acute Kidney Injury.

DETAILED DESCRIPTION:
After approval from the local Bioethics Committee of the Medical University of Gdańsk in Poland, the study was carried out between February 2019 and February 2020 among 32 patients admitted to ICU. There was no need to obtain written consent from the patients since the study was observational with no therapeutic intervention and decisional incapacity caused either by sedative drugs or severe condition of the patient.

Patients with acute kidney injury and indications for initiation of continuous renal replacement therapy (CRRT) were included to this study irrespective of their gender, race and age. Exclusion criteria were patients with previous end-stage chronic kidney disease treated with dialysis.

After decision to implement CRRT the serial blood samples were collected into two red-top tube (no anticoagulant or preservative) before initiation of CRRT and at 1,2,3,6,9,12,15,18-day following. Last samples were collected 3 days after the end of CRRT. Level of TSH, fT3 and fT4 were checked from the first tube after collecting the blood. Second tube was kept frozen until levels of TRH, TT3, TT4, rT3 could be measured. In all the patients high-dose continuous veno-venous hemodiafiltration (CVVHDF) with citrate anticoagulation was performed. Blood flow and dialysis dosage were the same for every patient depending on their weight. The weight was rounded up or down and patients were assigned to the nearest group.

ELIGIBILITY:
Inclusion Criteria:

Patients with acute kidney injury and indications for initiation of continuous renal replacement therapy (CRRT)

Exclusion Criteria:

Exclusion criteria were patients with previous end-stage chronic kidney disease treated with dialysis or with history of hypothyroidism.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with acute kidney injury and indications for continuous renal replacement therapy without pre-existing end-stage chronic kidney disease or hypothyroidism.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
blood concentrations of thyroid hormones | Samples were collected up to 1 hour before initiation and after 24, 48, 72, 144, 216 hours after initiation of CRRT. Last sample was collected 72 hours after the end of CRRT.
  TSH, fT3, fT4, TRH, TT3, TT4, rT3

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdansk - Departament of Anesthesiology and Intensive Care, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
share only results